CLINICAL TRIAL: NCT05437952
Title: Metabolic and Molecular Responses Under the Effect of Taurine Supplementation With and Without Multicomponent Training in Elderly Women With Sarcopenic Obesity Using the Metabolomics Approach
Brief Title: Metabolic and Molecular Responses Under the Effect of Taurine Supplementation With and Without Multicomponent Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: taurine_training_metabolomics
Record Dates: First submitted 2022-06-16; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Sarcopenic Obesity
Keywords: Sarcopenic Obesity; Aging; Taurine; Multicomponent Training; Metabolomics
MeSH Terms: interventions — Taurine; Exercise; tau Proteins

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical trial
Who Masked: Participant, Investigator
Masking Description: The study will involve 60 elderly women with sarcopenic obesity who will be randomly distributed into 4 groups: 1) GPL, submitted to placebo supplementation (n=15); 2) GTAU, submitted to taurine supplementation (n=15); 3) GPL+EX, submitted to placebo supplementation associated with physical exercise (n=15) and 4) GTAU+EX, submitted to taurine supplementation associated with physical exercise (n=15).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Taurine and Exercise (Tau+Ex) (Experimental): Participants who will receive 3g of taurine supplementation associated with physical training in the period of 16 weeks.
  Interventions: Dietary Supplement: Taurine and Exercise (Tau+Ex)
- Placebo and Exercise (PL+Ex) (Experimental): Participants who will receive 3g of placebo supplementation associated with physical training in the period of 16 weeks.
  Interventions: Other: Placebo and Exercise (PL+Ex)
- Taurine (Tau) (Experimental): Participants who will receive 3g of taurine supplementation in the period of 16 weeks.
  Interventions: Dietary Supplement: Taurine (Tau)
- Placebo (PL) (Placebo Comparator): Participants who will receive 3g of placebo supplementation in the period of 16 weeks.
  Interventions: Other: Placebo (PL)

INTERVENTIONS:
Dietary Supplement: Taurine and Exercise (Tau+Ex) — Participants will receive 3g of taurine to be supplemented in the morning in single-dose capsules. The intervention will last 16 weeks.
  Pshysical exercise
  Participants will perform a multicomponent type workout that explores strength, aerobic and balance capacities with load progression every 15 days. The sessions will last 60 minutes each, being held three times a week with a day of rest in between. The intervention will last 16 weeks
  Arms: Taurine and Exercise (Tau+Ex)
Other: Placebo and Exercise (PL+Ex) — Participants will receive 3g of placebo to be supplemented in the morning in single-dose capsules. The intervention will last 16 weeks.
  Pshysical exercise
  Participants will perform a multicomponent type workout that explores strength, aerobic and balance capacities with load progression every 15 days. The sessions will last 60 minutes each, being held three times a week with a day of rest in between. The intervention will last 16 weeks.
  Arms: Placebo and Exercise (PL+Ex)
Dietary Supplement: Taurine (Tau) — Participants will receive 3g of taurine to be supplemented in the morning in single-dose capsules. The intervention will last 16 weeks.
  Arms: Taurine (Tau)
Other: Placebo (PL) — Participants will receive 3g of placebo to be supplemented in the morning in single-dose capsules. The intervention will last 16 weeks.
  Arms: Placebo (PL)

SUMMARY:
Sarcopenic obesity is characterized by a progressive decline in muscle mass and an increase in body fat, a condition especially present in the elderly. A significant improvement in metabolic parameters has been observed with the completion of taurine supplementation and also with the practice of physical exercise, but there are no studies associating the interventions mentioned above with the aim of analyzing the metabolic profile of elderly people with sarcopenic obesity. The metabolomics approach allows the study of a whole set of metabolites involved in a biological system. It is believed that taurine supplementation associated with physical exercise is capable of promoting positive contributions to the metabolic profile, investigated through a metabolomics approach. Therefore, the present study seeks to investigate whether taurine supplementation associated with exercise is able to promote contributions to the metabolic profile, through a metabolomics approach, in elderly women with sarcopenic obesity.

DETAILED DESCRIPTION:
Sarcopenic obesity is characterized by a progressive decline in muscle mass and an increase in body fat, a condition especially present in the elderly. A significant improvement in metabolic parameters has been observed with the completion of taurine supplementation and also with the practice of physical exercise, but there are no studies associating the interventions mentioned above with the aim of analyzing the metabolic profile of elderly people with sarcopenic obesity. The metabolomics approach allows the study of a whole set of metabolites involved in a biological system. It is believed that taurine supplementation associated with physical exercise is capable of promoting positive contributions to the metabolic profile, investigated through a metabolomics approach. The study will involve 60 elderly women with sarcopenic obesity who will be randomly distributed into 4 groups: 1) GPL, submitted to placebo supplementation (n=15); 2) GTAU, submitted to taurine supplementation (n=15); 3) GPL+EX, submitted to placebo supplementation associated with physical exercise (n=15) and 4) GTAU+EX, submitted to taurine supplementation associated with physical exercise (n=15). The interventions will take place for 16 weeks, collections and evaluations will be carried out pre and post-intervention of functional capacity testing, anthropometry, resting energy expenditure, biopsy of white adipose tissue for analysis of gene expression and blood collection for analysis of the plasma concentration of taurine and of the metabolomic profile. Body composition, and food consumption will be evaluated pre, during and post-intervention. The synergistic effects of the proposed intervention are expected to improve the metabolic parameters, regarding the profile anti-inflammatory, antioxidant, lipid metabolism, body composition, and functional physical capacity in elderly women with sarcopenic obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 40kg/m²;
* Appendicular lean mass below 15 kg;
* Dynamometry below the cutoff point adjusted for sex and BMI (less than or equal to 21kg);
* "Sit and stand" test below the cut-off point adjusted for the age group, considering the number of repetitions in 30 seconds;
* Present medical certificate to perform physical exercise

Exclusion Criteria:

* alcoholics
* smokers;
* with any disease that prevents the practice of physical activity;
* medical impediment to the practice of physical exercise throughout the study;
* infectious diseases;
* coronary diseases;
* chronic kidney diseases;
* undergoing nutritional monitoring or weight loss treatment;
* score ≤13 for cognitive screening on the Mini-Mental State Examination (MMSE), suggested by Bertolucci et al. (1994).

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Metabolomic Profile | 16 weeks
  Changes in metabolites and lipids of the biological sample investigated through the metabolomics approach.

SECONDARY OUTCOMES:
Gene expressions in the subcutaneous white adipose tissue (scWAT). RNA (mRNA) levels of infammatory gene markers. | 16 weeks
  Changes in the expression of genes related to the inflammatory process that will be analyzed: C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-10 (IL-10), interleukin-15 (IL-15), necrosis factor tumor-α (TNF-α), nuclear factor-κβ (NFκβ) and adiponectin (ADIPOQ).
Gene expressions in the subcutaneous white adipose tissue (scWAT). RNA (mRNA) levels of oxidative stress genes markers. | 16 weeks
  Changes in the expression of genes related to oxidative stress that will be analyzed: superoxide dismutase (SOD1), glutathione peroxidase (GPx1) and catalase (CAT).
Gene expressions in the subcutaneous white adipose tissue (scWAT). RNA (mRNA) levels of lipid oxidation genes markers. | 16 weeks
  Changes expression of genes related to the lipid oxidation process that will be analyzed: sirtuin-1 (SIRT-1), forkhead O 1 (FOXO1), peroxisome proliferator 1 alpha (PGC-1α), peroxisomal proliferator alpha type (PPARα).
Functional ability tests: Six-minute walk test (minutes) | 16 weeks
  Changes in functional capacity assessed by: six-minute walk test.
Functional ability tests: forearm flexion test (seconds) | 16 weeks
  Changes in functional capacity assessed by: forearm flexion test.
Functional ability tests: muscle strength (dynamometer) - highest peak force (KGF) | 16 weeks
  Changes in functional capacity assessed by: muscle strength (dynamometer).
Functional ability tests: chair sit-up test. (seconds) | 16 weeks
  Changes in functional capacity assessed by: chair sit-up test.
Indirect calorimetry assessment | 16 weeks
  Changes in resting metabolic rate (RMR) evaluated pre and post intervention by indirect calorimetry.
Body composition changes (%) | 16 weeks
  Changes in % fat-free mass and fat mass evaluated pre, during and post intervention by iDEXA.
Anthropometric measurements (Body weight) | 16 weeks
  Changes in body weight (kilograms - Kg) pre and post intervention.
Anthropometric - height assessment (meters) | 16 weeks
  Height measured in meters
Anthropometric measurements (Circumferences) | 16 weeks
  Changes in waist, abdominal, and hip circumferences (centimeters) evaluated pre and post intervention.
Others changes in metabolic parameters | 16 weeks
  Changes in total cholesterol, triglycerides, HDL-cholesterol and LDL-c, fasting glucose and insulin sensitivity evaluated pre and post intervention.
Food Intake changes | 16 weeks
  Changes in food consumption. It will be evaluated through 24-hour food records. The professional software Dietbox will be used to evaluate the total consumption of energy and macronutrients. Evaluated pre, during and post intervention.
Changes in Plasma Taurine Concentration | 16 weeks
  Changes in Plasma Taurine Concentration. Plasma taurine will be determined by high performance liquid chromatography (HPLC).

CONTACTS AND LOCATIONS:
Overall Officials: Ellen C de Freitas, Ph.D., Principal Investigator — University of São Paulo, School of Physical Education and Sports of Ribeirão Preto

IPD SHARING:
Plan to Share IPD: No